CLINICAL TRIAL: NCT05657223
Title: Attending Physician, Division of Periodontics, Department of Dentistry, Kaohsiung Medical University Hospital, Kaohsiung
Brief Title: Factors Associated With the Complexity of Dental Implant Surgery After Alveolar Ridge Preservation: A Retrospective Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(I)-20210023
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: the Complexity of Implant Surgery
Keywords: periodontitis, alveolar ridge preservation, implant surgery.
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alcohol consumption, tooth position, and periodontitis-related tooth extraction affect the complexity of subsequent implant surgery after alveolar ridge preservation.

DETAILED DESCRIPTION:
Materials and methods We retrospectively analyzed the dentition of 165 alveolar ridge preservation sites in 116 patients. The bone width at three different vertical levels was measured on cone beam computed tomography images, and a comparison of bone regeneration requirements for subsequent dental implant surgery was performed for different socket types.

ELIGIBILITY:
Inclusion Criteria:

* teeth extraction in the premolar and molar regions, who underwent flapless tooth extraction with alveolat ridge preservation (ARP) and filling with freeze-dried bone allograft (FDBA) and platelet-rich fibrin (PRF), who underwent cone beam computed tomography (CBCT) followed by dental implant surgery after tooth extraction, and with adequate oral hygiene

Exclusion Criteria:

* untreated periodontitis, systemic disease, or the of medication that influences bone metabolism

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Of 165 sites, dental implant surgery was performed at 156 sites. A total of 72 damaged sockets and 93 intact sockets were included.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Alveolar bone width | 4~6 months

REFERENCES:
- [Derived] Hu KF, Chou YH, Lan CC, Ho PS, Liu PF, Tseng CJ. Greater bone regeneration required for implants following periodontal extraction: a retrospective cross-sectional study. BMC Oral Health. 2025 Apr 18;25(1):586. doi: 10.1186/s12903-025-05687-y. PMID 40251510